CLINICAL TRIAL: NCT02440867
Title: Treating Social Cognition Impairments in Patients With Schizophrenia With Repetitive Transcranial Magnetic Stimulation (Theta-Burst; TBS); a Pilot Study
Brief Title: Treating Social Cognition With Theta Burst Stimulation; a Pilot Sudy
Acronym: PilotTMS-COG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-A00839-38
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Social Cognition in Patients With Schizophrenia
Keywords: theta burst stimulation; Social Cognition; MRSI; Schizophrenia; transcranial magnetic stimulation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy subjects (No Intervention): Multimodal imaging data acquisitions Clinical data acquisitions
- TBS-MPC (Experimental): * Intervention with active TBS aiming Medial Prefrontal Cortex in 6 patients with schizophrenia
  * Baseline: Multimodal imaging data acquisitions; Clinical data acquisitions; P50 acquisition
  * Endpoint: Multimodal imaging data acquisitions; Clinical data acquisitions; P50 acquisition
  * Continuous actimetry acquisition
  Interventions: Device: Active TBS
- TBS-CPDLF (Active Comparator): * Intervention with active TBS aiming Dorsolateral Prefrontal Cortex in 6 patients with schizophrenia
  * Baseline: Multimodal imaging data acquisitions; Clinical data acquisitions; P50 acquisition
  * Endpoint: Multimodal imaging data acquisitions; Clinical data acquisitions; P50 acquisition
  * Continuous actimetry acquisition
  Interventions: Device: Active TBS
- TBS-Sham (Sham Comparator): * Intervention with Sham TBS in 8 patients with schizophrenia
  * Baseline: Multimodal imaging data acquisitions; Clinical data acquisitions; P50 acquisition
  * Endpoint: Multimodal imaging data acquisitions; Clinical data acquisitions; P50 acquisition
  * Continuous actimetry acquisition
  Interventions: Device: Sham TBS

INTERVENTIONS:
Device: Active TBS — Non-invasive transcranial magnetic stimulation inducing changes in cortical excitability depending on the cortical target (except for sham stimulation)
  Arms: TBS-CPDLF; TBS-MPC
Device: Sham TBS — Sham stimulation
  Arms: TBS-Sham

SUMMARY:
The purpose of the study is to test a new treatment of social cognition deficits in patients with schizophrenia or schizoaffective disorder by transcranial magnetic stimulation (theta-burst). The study will also identify clinical variables, cognitive and psychomotor most sensitive to treatment, to estimate the most sensitive treatment target, assess tolerance, to assess the impact of repetitive Transcranial Magnetic Stimulation (rTMS) on the brain a multimodal imaging study and compare the imaging variables (resting network, Diffusion Tensor Imaging, magnetic resonance spectroscopic imaging; MRSI) between patients before treatment and healthy subjects.

DETAILED DESCRIPTION:
The language understanding of other people is based on linguistic decoding mechanisms (phonological, semantic, syntactic ...) but also more on subtle mechanisms for the recognition of emotions and intentions. Interact with another one requires understanding its language but also to infer emotions and intentions. There are patients with schizophrenia suffering from social cognition disorders that impair social interactions; These patients often have difficulty in extracting the non-verbal emotional content of language and have difficulty inferring the thoughts and intentions of others. Recently, we have suggested a link between such deficits and the hypofunction of the medial prefrontal cortex.

Transcranial magnetic stimulation is a noninvasive neuromodulation technique that increases or decreases the focal cortical excitability depending on stimulation parameters. This technique is now commonly used as a therapeutic tool. It has been tried with some success in patients with schizophrenia in some indications:

* To reduce the auditory verbal hallucinations stimulating the temporal cortex
* More rarely, to reduce the negative symptoms stimulating the dorsolateral prefrontal cortex So far, the medial prefrontal cortex was not considered as a possible target as the scalp to cortex distance prevent from using conventional stimulation coils. Recently new coils have been developed that permit stimulation of deeper cortical regions.

We hypothesize that the use of transcranial magnetic stimulation with a theta burst intermittent protocol known to increase the cortical excitability and aiming the medial prefrontal cortex with a special antenna will improve social interaction capabilities of schizophrenic patients.

This ambitious and innovative assumption shall be first supported by a study of feasibility which is the subject of this trial.

Moreover, changes in the anatomical and functional connectivity, in brain metabolism and in cortical excitability will be observed after stimulation thanks to a multimodal imaging and the study of P50 wave.

In this pilot study, involving 20 patients, we plan to assess the social cognition deficits before and after 10 sessions of magnetic stimulation (2 sessions per day for 5 consecutive days) using a neuronavigation system and Magstim® stimulator. In order to assess the feasibility and specificity of the stimulation of medial prefrontal cortex (MPC), the effects of this treatment will be compared to the effects of the same treatment aiming the dorsolateral prefrontal cortex (DLPFC), also involved in aspects of negative symptoms of schizophrenia, and placebo effects induced by sham stimulation (using a sham coil). The recording of the P50 wave will be just before and after the 1st session and just after the last stimulation session. An MRI anatomical, functional and spectroscopic be performed before and 30 days after the treatment. A control group of twenty healthy subjects will perform the same MRI acquisitions.

ELIGIBILITY:
Inclusion Criteria:

* with a diagnosis of schizophrenia or schizoaffective disorder (DSM-IV MINI R)
* less than 20 years of disease duration
* Having signed a written informed consent
* LIS score > 15 or negative PANSS score > 15

Exclusion Criteria:

* Any change in psychotropic drugs (antidepressants, antipsychotics or mood stabilizers) during the two months preceding the inclusion
* Pregnant or breastfeeding women
* Subjects with a neurological condition or with epilepsy
* Subjects with a counter-indication to MRI or Transcranial stimulation (electronic or metal implants)
* Subjects that refuse to wear earplugs during MRI

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
V-LIS total score | change from baseline in V-LIS total score compared to 30 days after the end of the treatment

SECONDARY OUTCOMES:
GLX ratio | change in baseline GLX ratio measured in MRSI compared to 30 days after the end of the treatment
  GLX (= Glutamine + Glutamate) ratio are measured in the DLPFC and in the MPC
P50 wave amplitude | change in baseline P50 amplitude compared to immediately after the end of the treatment
Motor activity | change in baseline motor activity measured with an actimeter compared to 30 days after the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clément Nathou, MD, Principal Investigator — University Hospital, Caen
Locations (1):
- CHU de Caen - Centre Esquirol, Caen, France